CLINICAL TRIAL: NCT01399047
Title: Phase II, Randomized, Placebo Controlled Trial of the Safety and Tolerability of Mycophenolate in Children With Juvenile Neuronal Ceroid Lipofuscinosis
Brief Title: Cellcept for Treatment of Juvenile Neuronal Ceroid Lipofuscinosis
Acronym: JUMP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Batten Disease Support and Research Assocation (BDSRA) (Unknown)
Responsible Party: Principal Investigator, Erika Augustine, PI, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3908
Record Dates: First submitted 2011-07-05; First posted 2011-07-21 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Juvenile Neuronal Ceroid Lipofuscinosis
Keywords: Batten Disease
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate Mofetil (Active Comparator)
  Interventions: Drug: Mycophenolate mofetil
- Placebo liquid (Placebo Comparator)
  Interventions: Drug: Liquid Placebo

INTERVENTIONS:
Drug: Mycophenolate mofetil — The liquid dosage will be individualized, contingent upon the subject's weight. Subjects will receive 50% of the target dose (300mg/m2/dose BID) during Week 0-Week 2, then increase to the full dose (600mg/m2/dose BID) in Week 3, continuing at this dose through Week 8. Additionally, due to the risk of gastrointestinal disturbance (hemorrhage, ulcer), children will also receive prophylactic Prilosec (Omeprazole) for the duration of the study, during both the mycophenolate and placebo arms.
  Other Names: Cellcept
  Arms: Mycophenolate Mofetil
Drug: Liquid Placebo — The dosage will be individualized, contingent upon the subject's weight. Subjects will receive 50% of the target dose (300mg/m2/dose BID) during Week 0-Week 2, then increase to the full dose (600mg/m2/dose BID) in Week 3, continuing at this dose through Week 8. Additionally, due to the risk of gastrointestinal disturbance (hemorrhage, ulcer), children will also receive prophylactic Prilosec (omeprazole) for the duration of the study, during both the mycophenolate and placebo arms.
  Arms: Placebo liquid

SUMMARY:
The primary objective of this trial is to establish the safety and tolerability of short-term (8 weeks) administration of mycophenolate mofetil in ambulatory children with JNCL. The secondary objective is to gather preliminary evidence of the short-term (8 week) impact of mycophenolate mofetil on clinically relevant features of JNCL as measured by the Unified Batten Disease Rating Scale (UBDRS), including motor features, seizures, behavior, cognitive and functional measures.

Funding source-FDA Office of Orphan Product Development (OOPD).

DETAILED DESCRIPTION:
Juvenile Neuronal Ceroid Lipofuscinosis (JNCL) is a fatal disorder. Currently treatment is symptomatic. Thus, there is a real need to intervene and slow the progression of this disease. Preliminary data on genetic knock-down of the ability to mount an immune response in cln3-knockout mice is supportive of a strategy for treating JNCL with an immuno-suppressive agent. Many drugs with the ability to suppress the immune system are steroidal and deemed unsuitable for long-term administration to children. Mycophenolate mofetil (CellCept) is used as an immunosuppressive agent in allogenic transplants in pediatric patients and is therefore approved by the Food and Drug Administration (FDA) for pediatric use.

The study design is a double-blind, randomized, 22-week cross-over study of mycophenolate mofetil vs. placebo. After a 4-week washout period, subjects will undergo blinded crossover from active study drug to placebo or from placebo to active study drug.

Subjects and caregivers will be evaluated in person in the University of Rochester Batten Center (URBC) at screening/baseline, and at weeks 8, 12, and 20. In addition, subjects will be evaluated by their local clinician who is a formalized member of the research team. Such contacts will occur at Weeks 2, 4, 14, 16, and any unscheduled or early termination visits. There will also be regular telephone contact between the URBC and the local clinician.

We have selected the dosage currently FDA approved for use in children being treated for prophylaxis of renal transplant rejection.

ELIGIBILITY:
Inclusion Criteria:

* JNCL as determined by a characteristic clinical presentation and confirmatory genetic evidence.
* Able to walk 10 feet without assistance beyond that required due to vision impairment.
* Subjects with local treating clinician (pediatrician or neurologist) willing to conduct the trial according to the protocol, good clinical practice, and applicable regulations.
* Subjects with a parent/legal guardian willing to accompany them to all study visits, oversee study drug compliance, and monitor and report to local treating clinician/investigator and the URBC investigative personnel any signs of adversity.

Exclusion Criteria:

* Inability to tolerate oral administration of medications
* Concomitant medical condition, which, in the opinion of the local treating clinician, the parent(s)/guardian, or the URBC study investigator would place the child at greater than acceptable risk from: 1) travel by plane or car to the URBC on four occasions over the course of 22 weeks, 2) exposure to mycophenolate mofetil at protocol defined dosages for periods up to 8 weeks.
* Anticipated inability of the child (on the part of the investigator, parent/guardian, or URBC study personnel) to comply with the rigors of the protocol..
* Use of disallowed concomitant medications.
* Administration of immunosuppressive medications
* History of any prior exposure to mycophenolate mofetil
* History of hypersensitivity to mycophenolate mofetil, or any other component of the product
* History of frank gastrointestinal hemorrhage, ulceration, or melena
* White blood cell count < 3000/μL, absolute neutrophil count (ANC) < 1500/μL, hemoglobin < 10g/dL, or thrombocytopenia <100,000/μL.
* Abnormal liver function (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or bilirubin greater than 3 times the upper limit of normal)
* Pregnancy or vulnerability to engage in sexual intercourse based on report of the parent/guardian, judgment of the local treating clinician/investigator or judgment of the URBC study personnel.
* Positive Tuberculosis test
* Immunizations not up to date for age according to Centers for Disease Control guidelines

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2011-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika F Augustine, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Adams HR, Defendorf S, Vierhile A, Mink JW, Marshall FJ, Augustine EF. A novel, hybrid, single- and multi-site clinical trial design for CLN3 disease, an ultra-rare lysosomal storage disorder. Clin Trials. 2019 Oct;16(5):555-560. doi: 10.1177/1740774519855715. Epub 2019 Jun 11. PMID 31184505
- [Derived] Augustine EF, Adams HR, Mink JW. Clinical trials in rare disease: challenges and opportunities. J Child Neurol. 2013 Sep;28(9):1142-50. doi: 10.1177/0883073813495959. PMID 24014509

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Mycophenolate to Placebo Crossover: Subjects received one treatment period (8 weeks) of mycophenolate, then, after a 4-week washout, received one treatment period (8 weeks) of placebo, in a blinded manner.
- Group B: Placebo to Mycophenolate Crossover: Subjects received one treatment period (8 weeks) of placebo, then, after a 4-week washout, received one treatment period (8 weeks) of mycophenolate, in a blinded manner.
Period: Overall Study
Arm/Group | Group A: Mycophenolate to Placebo Crossover | Group B: Placebo to Mycophenolate Crossover
Started | 10 | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Mycophenolate to Placebo Crossover | Group B: Placebo to Mycophenolate Crossover | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.50 (5.99) | 14.78 (2.44) | 12.53 (5.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 7 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 9 | 8 | 17
  Race: More than one Race | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Tolerability - Number of Participants Who Completed Each Arm on Assigned Study Drug Dose
Description: The primary outcome measure is tolerability, defined as the completion of 8 weeks on the assigned dosage of study drug.
Time Frame: Baseline to 8 weeks
Population: All subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Mycophenolate: Includes data from all subjects while on mycophenolate, regardless of treatment order.
- Placebo: Includes data from all subjects while on placebo, regardless of treatment order.
Arm/Group | Mycophenolate | Placebo
Number analyzed (Participants) | 19 | 19
Participants | 17 | 19
Statistical Analysis 1: Comparison: Mycophenolate vs Placebo; The primary outcome variable was tolerability, defined as the proportion of subjects able to complete 8 weeks on the assigned treatment. Tolerability was compared among the treatment groups using Prescott's test. A 95% confidence interval was computed for the tolerability of mycophenolate, placebo, and their difference; Test type: Superiority or Other; p = 0.21, Prescott's test; Risk Difference (RD) = 0.105, 95% CI 2-sided [-0.033 to 0.243] — Mycophenolate was tolerated in 17/19 subjects (89.5%, 95% CI: 66.9% - 98.7%), while placebo was tolerated in 19/19 subjects (100%, 95% CI: 82.4% - 100%). The difference in tolerability rates was 10.5% (95% CI: -3.3% - 24.3%, p=0.21)

2. Secondary Outcome: Unified Batten Disease Rating Scale Physical Subscale Change
Description: The Unified Batten Disease Rating Scale (UBDRS) is a disease-specific clinical assessment. Motor impairment was measured by the physical subscale of the UBDRS with a range of 0-112 with zero indicating better outcome.
  The overall treatment effect was determined - mean difference in physical subscale change (Mycophenolate minus placebo periods) in outcome, adjusted for baseline value and period effects.
Time Frame: Baseline to 8 weeks
Population: All subjects who completed 8 weeks of the respective treatment arm assignment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mycophenolate: All data from subjects while on mycophenolate, regardless of treatment order.
- Placebo: All data from subjects while on placebo, regardless of treatment order.
Arm/Group | Mycophenolate | Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | -1.18 [-4.39 to 2.04] | 2.17 [-1.02 to 5.35]
Statistical Analysis 1: Comparison: Mycophenolate vs Placebo; Test type: Superiority or Other; p = 0.72, Prescott's test; Mean Difference (Net) = -0.69, 95% CI 2-sided [-4.67 to 3.28]

3. Secondary Outcome: Unified Batten Disease Rating Scale Seizure Subscale Change
Description: The Unified Batten Disease Rating Scale (UBDRS) is a disease-specific clinical assessment. Seizure severity was measured by the seizure subscale of the UBDRS with a range of 0-54 with zero indicating better outcome.
  The overall treatment effect was determined - mean difference in seizure subscale change (Mycophenolate minus placebo periods) in outcome, adjusted for baseline value and period effects.
Time Frame: Baseline to 8 weeks
Population: All subjects who completed 8 weeks of the respective treatment arm assignment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mycophenolate | Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | -0.24 [-1.15 to 0.68] | -1.44 [-3.03 to 0.14]
Statistical Analysis 1: Comparison: Mycophenolate; Test type: Superiority; p = 0.78, Prescott's test

4. Secondary Outcome: Unified Batten Disease Rating Scale Behavior Subscale Change
Description: The Unified Batten Disease Rating Scale (UBDRS) is a disease-specific clinical assessment. Mood and behavior severity was measured by the behavior subscale of the UBDRS with a range of 0-55 with zero indicating better outcome.
  The overall treatment effect was determined - mean difference in behavior subscale change (Mycophenolate minus placebo periods) in outcome, adjusted for baseline value and period effects.
Time Frame: Baseline to 8 weeks
Population: All subjects who completed 8 weeks of the respective treatment arm assignment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mycophenolate | Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | -1.28 [-4.12 to 1.56] | -0.37 [-2.94 to 2.20]
Statistical Analysis 1: Comparison: Mycophenolate; Test type: Superiority; p = 0.98, Prescott's test

5. Secondary Outcome: Unified Batten Disease Rating Scale Capability Subscale Change
Description: The Unified Batten Disease Rating Scale (UBDRS) is a disease-specific clinical assessment. Capability severity was measured by the capability subscale of the UBDRS with a range of 0-14 with higher scores indicating better outcome.
  The overall treatment effect was determined - mean difference in capability subscale change (Mycophenolate minus placebo periods) in outcome, adjusted for baseline value and period effects.
Time Frame: Baseline to 8 weeks
Population: All subjects who completed 8 weeks of the respective treatment arm assignment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mycophenolate | Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | 0.33 [-0.18 to 0.85] | 0.47 [-0.02 to 0.97]
Statistical Analysis 1: Comparison: Mycophenolate; Test type: Superiority; p = 0.26, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: Reporting of adverse events were sought at each encounter and were considered in the evaluation of each safety assessment (laboratory studies, electrophysiology).
Groups:
- Mycophenolate: Includes data from all subjects while on mycophenolate, regardless of order.
- Placebo: Includes data from all subjects while on placebo, regardless of order.
Arm/Group | Mycophenolate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19
Other Adverse Events (participants affected / at risk) | 14/19 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate (N=19) | Placebo (N=19)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate (N=19) | Placebo (N=19)
ECG Abnormality (Cardiac disorders) | 0 (0) | 1 (1)
Haemotympanum (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Weight decreased (Endocrine disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (8) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Strep pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Blood prolactin increased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 2 (2) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormality (Investigations) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Disorientation (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 0 (0) | 2 (2)
Movement disorder (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Abnormal behavior (Psychiatric disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 2 (2)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Perseveration (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes